CLINICAL TRIAL: NCT07314112
Title: Motivation, Learning and Decision Making in Changing Environments
Acronym: MOTILEARN
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital le Vinatier (Other)
Collaborators: INSERM U1208 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-A02725-42; VP2024-09 (Other: Hôpital Le Vinatier)
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Neurocognitive Model; Decision-Making
Keywords: Cognitive neurosciences; decision making; reward; cognitive psychology; fMRI

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Farming game: motivational fluctuation task: participants can gain points by engaging in some activities in the environment or just staying in one place. Throughout the experiment the level of reward for each patch will change to measure participants' sensitivity to different reward levels.
- Fastest Queue: prospective planning and learning task: participants observe two queues moving at different speeds shown to them in the middle of the screen. They need to decide which of two queues to stand in, and are asked about their beliefs about how fast individual queue members might get to the goal.
- Treasure hunt: sequential and incremental goal pursuit task: Participants need to decide between multiple goals to pursue framed as treasures in order to gain points. The treasures can be worth different amounts and the participant will be travelling to them at different speeds.

SUMMARY:
The main objective of this study is to develop a models of sequential decision-making, learning and motivation that includes emotions as driving forces of adaptive behaviour. Using functional magnetic resonance imaging (fMRI), the investigators will test the hypotheses that distinct parts of the prefrontal cortex play specific roles in naturalistic decision-making.

The main hypothesis is that distinct regions of the prefrontal cortex will be differentially involved in learning, motivation, and decision-making in naturalistic tasks. More specifically, the investigators hypothesise that by using a novel set of tasks they have designed in combination with fMRI, they can construct a neurocognitive model that explains how humans make adaptive decisions in dynamic and temporally extended reward environments.

A key region that the investigators believe will play a role in representing the internal and external parameters necessary for adaptive behaviours in the tasks is the anterior cingulate cortex. Depending on the task requirements, this region will further interact with other distinct prefrontal regions such as the frontal pole or dorsolateral prefrontal cortex.

Secondary hypotheses will also be investigated, specific to each specific task.

All data will be collected during a single visit lasting approximately 3.5 hours for each participant. Participants will perform a cognitive task inside the MRI scanner. Each participant will perform only one of the three possible cognitive conditions/tasks (Treasure Hunt, Fastest Queue, or Farm Game).

Each task is presented in the form of a video game played on a computer. Participants play a character who makes repeated choices. Participants are asked to try to collect as many points as possible within a limited time frame (Farm Game) or with limited trials (Fastest Queue and Treasure Hunt).

DETAILED DESCRIPTION:
Being able to make adaptive decisions and follow through on them is crucial for animals and humans alike. Although some simplifications of real-world environments are necessary for laboratories, previous studies have often removed an essential element of complexity: behaviour is often a sequence of choices, requiring planning, goal pursuit, and sustained motivation to achieve those goals. A comprehensive understanding of the brain functions at work and their cognitive, computational, and neural roles in these particular extended behaviours can only be achieved by examining the cognition and behaviour integrated into these extended temporal sequences.

In recent years, the investigators have addressed this challenge by developing a new neuroethological approach, made possible by advances in computational modelling, experimental design, brain recording and stimulation techniques. In this proposal, they have identified key cognitive processes related to the challenge of sequential and self-determined behaviours, behaviours enabled by the evolution of the prefrontal cortex, which underpins them through interactions with subcortical structures and associative cortical areas. To make this complexity manageable, they draw inspiration from several disciplines, including ecology, biology, psychology, and neuroscience. In this way, the investigators can identify the essential elements that enable complex adaptive behaviour in response to real-life challenges and build behavioural models around these processes.

For example, using this framework, our team challenged the notion that risk-taking propensity is a fixed characteristic in individuals. Instead, the investigators discovered that humans can flexibly modify the level of risk they are willing to take depending on the environment, particularly when searching for resources - in the same way that a bird close to starvation would take greater risks when searching for food.

An equally overlooked element of real-life decision-making is the interaction between emotions and decision-making, particularly during prolonged learning and decision-making over time, despite its potential relevance for understanding state-dependent decision-making, individual differences, and clinical disorders .

The current project aims to address three specific aspects of resource search. First, ecological environments often require advance planning, taking into account not only future opportunities present in the environment, but also behavioural tendencies and biases specific to the individual (e.g., the ability to exploit these future opportunities) in order to pursue long-term goals.

Second, in these situations, it is important to use any knowledge of the direction in which an environment is changing to plan ahead and use specific evaluation mechanisms to assess the gradual pursuit and abandonment of goals. Thirdly, at the same time, as these environments require consideration of a longer-term commitment, it is essential to understand how fluctuations in motivation can help or hinder these processes.

All data will be collected during a single visit for each participant. For each of the three tasks, the procedure will be the same; only the cognitive task performed will differ.

Part 1 of the visit = Setup, explanation of the study, verification of inclusion and non-inclusion criteria, and signing of consent.

Then, participants will practice the cognitive task. Part 2 of the visit : MRI session (cognitive task + structural MRI + functional MRI + physiological measurements).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45
* Fluent in French (reading and speaking)
* Membership or entitlement to a social security plan
* Have given written, informed consent to take part in the study
* Normal or corrected-to-normal vision
* Right-handed
* Body mass index (BMI) between 18.5 and 30

Non-inclusion Criteria:

* contraindication to MRI: pacemaker, heart battery, cardiac defibrillator, certain heart valves or neurosurgical clips, cochlear implant, implanted automated injection systems (insulin pump), intraocular metal projectiles, people who work or have worked with metals (excluding X-rays prior to MRI).
* under guardianship or curatorship or deprived of their liberty
* Participating in a clinical trial or in a period of exclusion from a previous clinical trial
* Breast-feeding or pregnant women
* claustrophobia
* Neurological disorder or severe chronic illness (diabetes, heart, kidney, lung or liver disease, inflammatory disease, psychiatric illness, etc.).
* The participant does not wish to be informed of any abnormalities detected during the MRI examination.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Functional brain activity | baseline
  Brain activity will be indirectly measured using the BOLD (blood-oxygen-level dependent) signal to test the neural correlates of our key task variables extracted using our cognitive models to infer potential neural mechanisms in our neurocognitive model.

SECONDARY OUTCOMES:
Decisions on the Farming game | baseline
  The cognitive model of goal pursuit will be used to construct regressors that represent the different motivations for goal abandonment (specifically frustration, temptation, and avoidance). Significant correlations between these model regressors voxel-by-voxel will be tested in a mass univariate manner.
Decisions on the Fastest Queue task | Baseline
  The cognitive model of reward tendencies will be used to construct regressors that represent the use of reward tendency information. The significant correlations between these model regressors will be tested voxel-by-voxel in a mass univariate manner.
Decisions on the Treasure Hunt Game | Baseline
  The cognitive model of motivation and vigor will be used to construct regressors that represent the participant's emotional and motivational state. Significant correlations between these model regressors will be tested voxel by voxel in a mass univariate manner.

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kolling, PhD, Principal Investigator — INSERM U1208, Ecological Cognition and Computation Team
Locations (1):
- INSERM, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided